CLINICAL TRIAL: NCT07306559
Title: A Phase I Study to Determine the Safety and Tolerability of BI 3820768 in Patients With Advanced Relapsed or Refractory Germ Cell Tumours, Endometrial Cancer, or Ovarian Cancer
Brief Title: A Study to Test How Well Different Doses of BI 3820768 Are Tolerated by People With Advanced Cancer (Solid Tumours)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2001-0001; 2025-522913-45-00 (Registry Identifier: CTIS (EU)); U1111-1324-5961 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Advanced Relapsed or Refractory Germ Cell Tumours; Advanced Relapsed or Refractory Endometrial Cancer; Advanced Relapsed or Refractory Ovarian Cancer
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: BI 3820768 (Experimental)
  Interventions: Drug: BI 3820768
- Part 2: BI 3820768 (Experimental)
  Interventions: Drug: BI 3820768

INTERVENTIONS:
Drug: BI 3820768 — BI 3820768

SUMMARY:
This study is open to adults with advanced germ cell tumours, endometrial cancer, or ovarian cancer whose previous treatments were not successful. People can join the study if they have no remaining treatment options or if standard therapy is not suitable. The purpose of this study is to test increasing doses of BI 3820768 to find a dose that people with these types of cancer can tolerate and that may make tumours shrink. BI 3820768 is a type of treatment that may help the immune system fight cancer. This is the first time BI 3820768 is being tested in humans.

The study has 2 parts based on the way BI 3820768 is given. Depending on when participants join the study, they will receive BI 3820768 through one of two ways to inject the study medicine. All participants receive the study medicine. The medicine is given as an injection once a week for 2 cycles of 3 weeks each, followed by doses every 3 weeks.

Participants are in the study for up to 3 years if they are benefiting from the treatment. During this time, they visit the study site regularly, and some visits will require overnight stays. Doctors will regularly check the size of the tumour and whether it has spread. Researchers want to find the highest dose of BI 3820768 that participants can tolerate by looking at the number of participants with certain severe health problems. The doctors also regularly check participants' health, take blood samples, and note any unwanted effects.

ELIGIBILITY:
Inclusion criteria :

1. Patient must be ≥18 years of age and at least at the legal age of consent in countries where it is older than 18 years at the time of signature on the informed consent forms (ICFs).
2. For patients with endometrial cancer (EC) and ovarian cancer (OVC), signed and dated written ICF1 for target testing.
3. Signed and dated ICF2 for all patients describing the study in accordance with International Council on Harmonisation Good Clinical Practice (ICH-GCP) and local legislation prior to any trial-specific procedures, sampling, or analyses.
4. Prior to Screening Visit 02, confirmed target-positivity for EC and OVC based on central laboratory testing of tumour tissue sample.
5. Patients with a histologically or cytologically confirmed diagnosis of germ cell tumour (GCT), EC, or OVC.
6. Patients with advanced, relapsed/refractory (r/r) GCT, EC, or OVC.
7. Patients with disease progression despite conventional treatment, intolerant to or not a candidate for conventional treatment, who have exhausted all established treatment options.
8. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Further inclusion criteria apply.

Exclusion criteria:

1. Patient with a history of a major surgery within 28 days prior to the first dose of BI 3820768 (major according to the Investigator's and/or Sponsor's assessment).
2. Previous or concomitant malignancies other than the one treated in this trial within the past 3 years except:

   1. Effectively treated non-melanoma skin cancers
   2. Effectively treated carcinoma in situ of the cervix
   3. Effectively treated ductal carcinoma in situ
   4. Other effectively treated malignancy that is considered cured by local treatment
3. Patient with known leptomeningeal disease or spinal cord compression due to disease.
4. Presence of any infection requiring systemic antimicrobial treatment within 7 days prior to the first dose of trial medication. Patients who have any clinical signs of infection (e.g. fever or leukocytosis) within 48 h prior to the first dose of trial medication are not eligible.
5. Patients with Hepatitis-C-Virus (HCV) infection, defined as:

   1. Currently receiving curative antiviral treatment for HCV infection, and/or
   2. HCV viral load is above the limit of quantification (HCV RNA positive).
6. Patients with active hepatitis B virus (HBV) infection (chronic or acute); defined as having a positive hepatitis B surface antigen (HBsAg), and HBsAg test at screening.
7. Patient with past HBV infection or resolved HBV infection (defined as the presence of hepatitis B core antibody (HBcAb) and absence of HbsAg) are eligible. HBV DNA must be obtained in these patients prior study start.

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2029-04-21 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment-emergent AEs | up to 3 years.
  AEs=Adverse Events
Occurrence of DLT(s) | up to 3 years.
  DLT(s)=Dose Limiting Toxicities

SECONDARY OUTCOMES:
Objective response (OR) | up to 3 years.
  Defined as the best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), where Best overall response (BOR) is determined according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
Maximum measured plasma concentration of BI 3820768 after the first administration | up to 24 hours.
Maximum measured plasma concentration of BI 3820768 after multiple administrations | up to 3 years.
Area under the concentration-time curve of BI 3820768 after the first administration | up to 24 hours.
Area under the concentration-time curve of BI 3820768 after multiple administrations | up to 3 years.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (3):
  - Valkyrie Clinical Trials, Los Angeles, California
  - Indiana University, Indianapolis, Indiana
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
- France (2):
  - INS Paoli-Calmettes, Marseille
  - INS Gustave Roussy, Villejuif
- Germany (2):
  - Klinikum der Universität München AÖR, München
  - Universitätsklinikum Würzburg AÖR, Würzburg
- Japan (2):
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - Japanese Foundation for Cancer Research, Tokyo, Koto-ku
- Spain (2):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Clínica Universidad de Navarra - Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com